CLINICAL TRIAL: NCT00000859
Title: A Randomized Trial of the Efficacy and Safety of a Strategy of Starting With Nelfinavir Versus Ritonavir Added to Background Antiretroviral (AR) Nucleoside Therapy in HIV-Infected Individuals With CD4+ Cell Counts Less Than or Equal to 200/mm3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 042; 11592 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Resistance; Drug Therapy, Combination; HIV Protease Inhibitors; CD4 Lymphocyte Count; Ritonavir; Indinavir; Disease Progression; RNA, Viral; Genotype; Nelfinavir; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Indinavir; Ritonavir; Nelfinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Nelfinavir mesylate

SUMMARY:
To compare nelfinavir (NFV) with ritonavir (RTV) for delaying disease progression or death in HIV-infected patients with CD4+ cell counts less than 100 cells/mm3 [AS PER AMENDMENT 3/11/98: less than or equal to 200 cells/mm3]. To compare NFV with RTV for the development of adverse events and for rates of permanent discontinuation of study medication.

[AS PER AMENDMENT 10/02/97: To compare by intention-to-treat analysis for disease progression, including death, the following two regimens: NFV plus background combination antiretroviral (AR) therapy followed by indinavir (IDV) or RTV in the event of significant intolerance; and RTV plus AR therapy followed by IDV, then NFV, in the event of significant intolerance.] [AS PER AMENDMENT 3/11/98: SUBSTUDY CPCRA 045: To determine the relative rates of emergence of HIV-1 resistance and to compare changes in plasma HIV RNA levels and CD4+ cell counts in a sample of patients with CD4+ cell counts <= 200/mm3 who are enrolled in protocol CPCRA 042.] AR therapy is rapidly becoming the standard of care for the treatment of HIV infection. AR therapy provides the best opportunity for maximizing viral suppression, reducing toxicity and delaying the emergence of resistant strains. The newest class of AR agents, the HIV protease inhibitors, exhibits the most potent anti-HIV effects described to date. This study will compare 2 protease inhibitors, NFV and RTV for efficacy and safety in a population with advanced HIV disease, who are taking various background nucleoside therapies.

DETAILED DESCRIPTION:
AR therapy is rapidly becoming the standard of care for the treatment of HIV infection. AR therapy provides the best opportunity for maximizing viral suppression, reducing toxicity and delaying the emergence of resistant strains. The newest class of AR agents, the HIV protease inhibitors, exhibits the most potent anti-HIV effects described to date. This study will compare 2 protease inhibitors, NFV and RTV for efficacy and safety in a population with advanced HIV disease, who are taking various background nucleoside therapies.

Eligible patients will be randomized either to NFV plus background AR nucleoside therapy or to RTV plus background AR nucleoside therapy. Background AR therapy may also be no background therapy, although use of protease inhibitors as monotherapy is not recommended unless there is no alternative. Patients will be allowed to cross over to the alternate protease inhibitor if they reach a primary study endpoint. Data will be collected every 4 months.

[AS PER AMENDMENT 10/2/97: Patients assigned to the NFV arm who develop a significant intolerance may switch to RTV or IDV; those assigned to the RTV arm who develop a significant intolerance are encouraged to switch to IDV (NFV allowed if IDV contraindicated). Switchover for intolerance is strongly discouraged during the first 4 weeks of follow-up. Patients initially assigned to NFV therapy who experience disease progression may switch to RTV; if RTV is not tolerated, patients may switch to IDV. Because of the cross-resistance between RTV and IDV, patients who progress on RTV should switch to NFV.] [AS PER AMENDMENT 12/15/98: Patients originally assigned to NFV who experience poor virologic control or disease progression should change to RTV or IDV or enroll in the PIP protocol (CPCRA 057). Conversely, patients originally assigned to RTV should change to NFV or enroll in the PIP protocol (such patients continue to be followed on this study). Because of cross-resistance between RTV and IDV, change from RTV to IDV is discouraged. Determination of poor virologic control or disease progression is at the discretion of the patient's clinician. Change in background antiretroviral therapy should occur at the same time that the protease inhibitor is changed for poor virologic control or progression; the choice of new background antiretroviral agents is at the discretion of the clinician.] Randomization is stratified by clinical site.] [AS PER AMENDMENT 3/11/98: SUBSTUDY CPCRA 045: At least 600 patients (>= 400 from CPCRA sites and >= 200 from CTN sites) will be enrolled in the substudy. These patients will have a plasma sample collected for HIV RNA and genotypic resistance within 30 days prior to randomization, at the 1-month visit, and at the q-4-month study visits thereafter until the end of the study. CD4+ cell counts will be done at the 1-month visit and at the q-4-month study visits until the end of the study. A subset of patients will also have immunophenotyping of CD4+ and CD8+ cell TCR V-beta clones carried out before and during treatment. Another subset of patients at selected sites will have viral cultures performed for phenotypic drug sensitivity testing.

Initially, specimens for 50 randomly chosen patients in the group originally assigned RTV will be identified for resistance testing. Of this group, specimens for those who have received RTV/IDV for more than 1 month will be analyzed for genotypic resistance to obtain an estimate of the rate of resistance development and to estimate the risk of disease progression associated with resistance to RTV/ZDV. Based on these estimates, determination will be made of the total number of patients and specimens in both treatment groups in order to address the primary objective of comparing genotypic resistance in the two groups.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

* Background AR nucleoside therapy is required, although background AR therapy may also be no background therapy. However, the use of protease inhibitors is not recommended as monotherapy unless there is no other alternative. Therefore, patients who are not on AR treatment may be enrolled at the discretion of the clinician.

Allowed:

* Saquinavir.

Patients must have:

* Documented HIV infection.
* A CD4+ cell count <= 100/mm3 within 3 months prior to the study. [AS PER AMENDMENT 3/11/98: CD4+ cell count <= 200/mm3 any time prior to entry].
* Parental consent if patient is < 18 years old.

Prior Medication:

Allowed:

* Saquinavir (SQV).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Stage 2 or greater AIDS dementia complex.
* [AS PER AMENDMENT 10/2/97: Any acute disease or condition that would, in the physician's judgement, contraindicate starting NFV or RTV.]
* Known hypersensitivity to RTV or any of its ingredients (for patients assigned to RTV therapy).

Concurrent Medication:

Excluded:

* Concomitant use of protease inhibitors.
* Concomitant treatments that cannot be discontinued, and in the physician's judgement, should not be taken with NFV or RTV.

AS PER AMENDMENT 10/2/97:

* For patients randomized to NFV:
* Concomitant therapy with terfenadine, astemizole, cisapride, triazolam, midazolam, ergot derivatives, amiodarone, quinidine, or rifampin.

For patients randomized to IDV:

* Concomitant therapy with terfenadine, astemizole, cisapride, triazolam, midazolam, and rifampin.

Patients with any of the following prior symptoms are excluded:

AS PER AMENDMENT 10/2/97:

* History of clinically significant hypersensitivity reaction to any component of NFV tablets (for patients assigned to NFV therapy).

Prior Medication:

Excluded:

* Prior use of protease inhibitors except SQV.

[AS PER AMENDMENT 10/2/97:

* Prior use of IDV for more than 4 weeks or other protease inhibitors (except SQV) for any prior duration.]

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300
Dates: Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perez G, Study Chair; MacArthur R, Study Chair
Locations (44):
- United States (32):
  - Community Consortium / UCSF, San Francisco, California
  - Community Consortium of San Francisco, San Francisco, California
  - Denver Community Program for Clinical Research on AIDS, Denver, Colorado
  - Denver CPCRA / Denver Pub Hlth / Rocky Mt Cancer Ctr Aurora, Denver, Colorado
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Infectious Disease Physicians / Northern Virginia, Washington D.C., District of Columbia
  - Timothy A Price, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Louisiana Community AIDS Research Program, New Orleans, Louisiana
  - Baltimore TRIALS, Baltimore, Maryland
  - Westat / NICHD, Rockville, Maryland
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Wayne State Univ / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Mercer Area Early Intervention Services, Camden, New Jersey
  - Southern New Jersey AIDS Clinical Trials, Camden, New Jersey
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - New Jersey Community Research Initiative, Newark, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research - New Mexico, Albuquerque, New Mexico
  - Partners Research, Albuquerque, New Mexico
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Harlem AIDS Treatment Group, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Saint Joseph's Hosp, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia
- Canada (12):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Saint Joseph's Hosp, London, Ontario
  - Ottawa Gen Hosp, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Gen Hosp, Toronto, Ontario
  - Wellesley Hosp, Toronto, Ontario
  - Hotel - Dieu de Montreal, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - SMBD-Jewish Gen Hosp, Montreal, Quebec
  - Centre De Recherche En Infectiologie, Ste-Foy, Quebec
  - Royal Univ Hosp, Saskatoon, Saskatchewan

REFERENCES:
- [Background] MacArthur RD, Perez G, Walmsley S, Baxter J, Neaton J, Wentworth D. CD4 cell count is a better predictor of disease progression than HIV RNA level in persons with advanced HIV infection on highly active antiretroviral therapy. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 203)
- [Result] Perez G, MacArthur RD, Walmsley S, Baxter JA, Mullin C, Neaton JD; Terry Beirn Community Programs for Clinical Research on AIDS; Canadian Trials Network. A randomized clinical trial comparing nelfinavir and ritonavir in patients with advanced HIV disease (CPCRA 042/CTN 102). HIV Clin Trials. 2004 Jan-Feb;5(1):7-18. doi: 10.1310/N11F-NK93-MUMR-A1VV. PMID 15002082
- [Result] MacArthur RD, Perez G, Walmsley S, Baxter JD, Mullin CM, Neaton JD; Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA) 042/045; Canadian HIV Trials Network (CTN) 102 Protocol Teams. Comparison of prognostic importance of latest CD4+ cell count and HIV RNA levels in patients with advanced HIV infection on highly active antiretroviral therapy. HIV Clin Trials. 2005 May-Jun;6(3):127-35. doi: 10.1310/A9B9-RQD7-U8KA-503U. PMID 16192247